CLINICAL TRIAL: NCT02017639
Title: A Multi-center, Open-label, 2-treatment, Single-sequence Clinical Study to Evaluate the Effects of a Single 200 mg Subcutaneous Injection of Sarilumab on the Pharmacokinetics of a Single 40 mg Oral Dose of Simvastatin, With Optional 1-year Extension of Open Label Treatment of Sarilumab, in Patients With Rheumatoid Arthritis
Brief Title: Sarilumab Effect on the Pharmacokinetics of Simvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: INT12684; U1111-1140-5082 (Other: UTN)
Record Dates: First submitted 2013-12-02; First posted 2013-12-23 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sarilumab SAR153191 (REGN88) (Experimental): Single dose of simvastatin before and after sarilumab administration
  Interventions: Drug: sarilumab SAR153191 (REGN88); Drug: simvastatin

INTERVENTIONS:
Drug: sarilumab SAR153191 (REGN88) — Pharmaceutical form:Prefilled syringe of sarilumab solution Route of administration: Subcutaneous injection
Drug: simvastatin — Pharmaceutical form:Film-coated 20 mg Tablet Route of administration: oral

SUMMARY:
Primary Objective:

To evaluate the effect of a single 200 mg subcutaneous injection of sarilumab on the pharmacokinetics of simvastatin in patients with rheumatoid arthritis

Secondary Objective:

To describe the safety and efficacy (exploratory) of sarilumab

DETAILED DESCRIPTION:
The duration of the entire study per patient completing both Parts A and B is expected to be approximately 58 weeks (not including Screening).

ELIGIBILITY:
Inclusion criteria:

Male or female, between 18 and 75 years of age, inclusive. Body weight between 50.0 and 120.0 kg, inclusive, if male, and between 40.0 and 110.0 kg, inclusive, if female.

Diagnosis of RA, according to the ACR/European League against Rheumatism (EULAR) 2010 Rheumatoid Arthritis Classification Criteria with ≥ 3 months disease duration, ACR Class I-III functional status, based on 1991 revised criteria (Appendix B, 5). Moderate-to-severely active RA, defined as:

o high sensitivity C-reactive protein (hs-CRP) ≥ 6 mg/L

Laboratory parameters within the normal range (or defined screening threshold for the Investigator site), unless the Investigator considers an abnormality to be clinically irrelevant for RA patients; however following lab values must be met:

* Hemoglobin >8.5 g/dL
* White blood cells >3000/mm3
* Neutrophils >2000/mm3
* Platelet count >150 000 cells/mm3

Exclusion criteria:

Prior or current significant concomitant illness(es) that, according to Investigator's judgment, would adversely affect the patient's participation in the study.

Women of childbearing potential not protected by highly-effective contraceptive method(s) of birth control (as defined in the informed consent form), and/or who are unwilling or unable to be tested for pregnancy.

Participation in any clinical research study that evaluated an investigational drug or therapy within 5 half-lives or 60 days of the Screening, whichever is longer.

Patients with active TB or a history of incompletely treated TB. History of chronic infection or active infection. History of, or current, autoimmune or inflammatory systemic or localized joint disease(s) other than RA.

A systemic hypersensitivity reaction, other than localized injection site reaction, to any biologic drug.

History or presence of drug or alcohol abuse. Prior or current interstitial lung disease diagnosed by high resolution computed tomography and/or lung biopsy with consistent findings on pulmonary function tests and corroborating clinical findings.

Prior or current history of malignancy, including lymphoproliferative diseases, other than adequately-treated carcinoma in-situ of the cervix, nonmetastatic squamous cell or basal cell carcinoma of the skin, within 5 years prior to the screening visit.

Uncontrolled diabetes mellitus, defined as glycosylated hemoglobin (HbA1c) ≥9% at the screening visit.

Current treatment with anti-TNF agents or other biologics. Current treatment with RA-directed biologic agents with non- TNF-α antagonist. Any contra-indications to simvastatin, according to the applicable labeling. Current treatment with a statin within 14 days before inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assessment of PK parameters - area under curve from zero time until the last measurable concentration (AUClast) and AUC for simvastatin | Day 1 of Period 1 and Day 8 of Period 2

SECONDARY OUTCOMES:
Assessment of additional PK parameters for simvastatin | Day 1 of Period 1 and Day 8 of Period 2
Assessment of additional PK parameters for simvastatin acid | Day 1 of Period 1 and Day 8 of Period 2
Safety assessment of sarilumab up to 1 year ) | From Day 1 of Period 1 up to a maximum of 1 year (week 58)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- United States (3):
  - Investigational Site Number 840002, Duncansville, Pennsylvania
  - Investigational Site Number 840003, Jackson, Tennessee
  - Investigational Site Number 840001, Dallas, Texas
- Investigational Site Number 498001, Chisinau, Moldova
- Investigational Site Number 410002, Seoul, South Korea

REFERENCES:
- [Derived] Lee EB, Daskalakis N, Xu C, Paccaly A, Miller B, Fleischmann R, Bodrug I, Kivitz A. Disease-Drug Interaction of Sarilumab and Simvastatin in Patients with Rheumatoid Arthritis. Clin Pharmacokinet. 2017 Jun;56(6):607-615. doi: 10.1007/s40262-016-0462-8. PMID 27722854